CLINICAL TRIAL: NCT05245604
Title: A Phase Ⅲ, Multicenter, Randomized, Double-blind, Active-controlled, Parallel Study of TJO-087 for Evaluating 32 Weeks Safety and Efficacy in Moderate to Severe Dry Eye Disease Patients
Brief Title: Evaluating the Efficacy and Safety of TJO-087 in Moderate to Severe Dry Eye Disease Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taejoon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TJO-087-301
Record Dates: First submitted 2022-02-08; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TJO-087 (Experimental)
  Interventions: Drug: TJO-087
- Cyclosporine 0.05% (Active Comparator)
  Interventions: Drug: Cyclosporine ophthalmic solution 0.05%

INTERVENTIONS:
Drug: TJO-087 — Cyclosporine ophthalmic nano-emulsion 0.08%, 1 drop once daily
  Arms: TJO-087
Drug: Cyclosporine ophthalmic solution 0.05% — Cyclosporine ophthalmic solution 0.05%, 1 drop twice/day
  Arms: Cyclosporine 0.05%

SUMMARY:
The purpose of this clinical study is to prove that the test drug (TJO-087) is not clinically inferior to the control drug after 32 weeks of administration to patients with suppressed tear production due to moderate or severe dry eye syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 20 or over
* Patients with moderate to severe dry eye
* Screening both eyes, the corrected visual acuity is 0.2 or more
* Written informed consent to participate in the trial

Exclusion Criteria:

* Screening visits within 2 weeks who treated with topical NSAIDs/hyaluronate sodium ophthalmic solutions
* Screening visits within 2 months the patients with systemic or ocular disorders affected the test results (ocular surgery, trauma, or disease)
* Intraocular pressure(IOP)> 25 mmHg
* Patient using or to use punctual plug within 1 months.
* Patients with contact lens.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2020-06-19 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Non-anesthetic Schirmer Test at Week 32 | Baseline and Week 32
  The Schirmer test without anesthesia was used to estimate tear flow stimulated reflexly by insertion of a filter paper strip into the conjunctival sac.

SECONDARY OUTCOMES:
Change From Baseline in Non-anesthetic Schirmer Test at Week 8, 16, 24 | Baseline, Week 8, 16 and 24
  The Schirmer test without anesthesia was used to estimate tear flow stimulated reflexly by insertion of a filter paper strip into the conjunctival sac.
Change From Baseline in Corneal Fluorescein Staining Score at Week 8, 16, 24 and 32 | Baseline, Week 8, 16, 24 and 32
  Change from Baseline in corneal staining of the worse eye using blue fluorescein staining procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Hyo Myung Kim, MD, PhD, Principal Investigator — Korea University Anam Hospital
Locations (1):
- Hyo Myung, Kim, Seoul, South Korea

REFERENCES:
- [Derived] Eom Y, Yoon KC, Kim HK, Song JS, Hyon JY, Kim HM. A Multicenter, Randomized, Double-Blind Evaluation of the Efficacy of TJO-087 Versus 0.05% Cyclosporine A in Moderate to Severe Dry Eye. J Ocul Pharmacol Ther. 2023 Jan-Feb;39(1):27-35. doi: 10.1089/jop.2022.0119. Epub 2022 Nov 24. PMID 36450107